CLINICAL TRIAL: NCT01159899
Title: Pilot Study of A One-Step Procedure for the Use of Autologous Bone Marrow Mesenchymal Stem Cells Stimulated by Proteins Scaffold to Heal Under Arthroscopy Full-Thickness Defects Articular Cartilage and Osteoarthrosis of the Knee.
Brief Title: Transplantation of Bone Marrow Stem Cells Stimulated by Proteins Scaffold to Heal Defects Articular Cartilage of the Knee
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Michel Assor, MD (Other)
Responsible Party: Sponsor-Investigator, Michel Assor, MD, Sponsor-Investigator, University of Marseille
Organization: University of Marseille (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MSC- AS3
Record Dates: First submitted 2010-07-06; First posted 2010-07-12 (Estimated); Last update posted 2013-01-08 (Estimated); Status verified 2013-01

CONDITIONS: Osteoarthritis; Knee Osteoarthritis; Osteochondritis Dissecans; Osteonecrosis
Keywords: Osteoarthritis; knee arthritis; Knee arthrosis; articular cartilage defects; osteochondral defects; mesenchymal stem cells; stem cells; cellules souches,; genou; arthrose genou; PRP platelet rich plasma; thérapie cellulaire; implantation cellules souches mésenchymateuses; régénération cartilage; cicatrisation ménisque; ligament; plasma riche plaquettaire; platelet rich plasma; stem cell; regrowt cartilage; cellules souches; PRP
MeSH Terms: conditions — Osteoarthritis; Osteoarthritis, Knee; Osteochondritis Dissecans; Osteonecrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Transplantation of Bone Marrow Stem Cells Activated in Knee Arthrosis — Transplantation of Activated Bone Marrow Stem Cells in Knee Arthrosis, under arthroscopy, in one-step procedure
  Other Names: mesenchymal stem cells; Knee Arthrosis; Knee osteochondral defect

SUMMARY:
The purpose of this pilot study is to investigate the efficacy and safety of autologous transplantation, under arthroscopy, of Bone Marrow Mesenchymal stem cells, using, with a cell separator, a fresh non-culture expanded Autologous Bone Marrow derived Mesenchymal Stem, mixed and activated with proteins scaffold in patient with Knee cartilage defects and osteoarthritis. Based on extensive preclinical investigations, the technology of using freshly isolated bone marrow mononuclear cells mixed with proteins seems safe and most effective for a one-step correction of cartilage defect and restoration of the osteochondral complex, because the same mixture can generate cartilage in the vasculature-free knee joint, and bone in the environment of bone defects.

DETAILED DESCRIPTION:
Before the implantation of the mesenchymal stem cells, a knee arthroscopy procedure is made for the debridement of the meniscal and cartilage lesions, with microperforation and abrasion, preparation of the osteochondral defect to receive the transplantation, patellar lateral release if necessary.

Then, the investigators use a fresh non-culture expanded autologous bone marrow derived mesenchymal mononuclear stem cells, stimulated with a protein matrix and mixed in a collagen hydroxyapatite scaffold. This cellular paste is transplanted in the prepared defect, under arthroscopy, with injection of platelet rich plasma.

ELIGIBILITY:
Inclusion Criteria:

* Active patients (30 to 75 years)
* A localized osteochondral defect of both condyle and/or tibia grade 4 (ICRS classification)
* with cartilage on the tibial surface no more than grade 3-4, of size < 3-4 cm2, with 3/4 of meniscus present.
* Stable knee ; previous ligament reconstruction, if stable
* A defect that is 1 - 4 cm2 or more, up to 6 cm2, located on the femoral condyle and /or less of 4 cm2 for tibial plate, and IKS score <75.
* Kissing lesions admitted
* Ability to understand and willingness to sign consent form

Exclusion Criteria:

* Patients younger than 30 years and older than 75 years
* Diffuse and advanced articular cartilage degeneration of the joint
* Axial malalignment, meniscal pathology, and ligamentous instability are relative contraindications that have to be dealt with primarily either concomitantly or before the transplantation during 1 of the 2 stages of the procedure. Refusal of the patient to address these conditions in presence of a cartilage lesion is a criterion for exclusion from the study, to avoid the impact of these knee pathologies on the final results
* Existing infection in or around the joint & lesions of infectious or oncologic etiology.
* Debilitated patients.
* Immunocompromised patients.
* Patients with autoimmune disorders & systemic inflammatory disease.
* Preoperative poor neurological or vascular status of the affected limb.
* Specific contraindications include the use of tobacco and medications that may impair cell proliferation, such as NSAIDs and immunosuppressive drugs. Patients must be nicotine-free (stop smoking) prior to the procedure, as studies have shown that the oxidative effect of smoking impairs cell function and subsequent healing.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2010-07; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
IKS, International Knee Score | 6 months
  measure assess of the knee function
IKS, International Knee Score | 1 year
  measure assess of the knee function

SECONDARY OUTCOMES:
KOOS, Knee Injury and Osteoarthritis Outcome Score | 6 months
  measure assess of the knee function and quality of the new cartilage
KOOS, Knee Injury and Osteoarthritis Outcome Score | 1 year
  measure assess of the knee function and quality of the new cartilage

CONTACTS AND LOCATIONS:
Overall Officials: Michel Assor, MD, Principal Investigator — Knee and Lower Limb Institute, Marseille, France; Shimon Slavin, MD, Study Director — The International Center for Cell Therapy & Cancer (ICTC), Tel Aviv, Israel
Locations (1):
- Knee and Lower Limb Institute, Dr Michel Assor, Marseille, France

REFERENCES:
- See also: knee stem cell procedures — http://cellulesouche-genou.blogspot.com
- See also: cell therapy and PRP — http://cellulesouches.org